CLINICAL TRIAL: NCT04097782
Title: Effects of Antenatal Education on Fear of Birth, Depression, Anxiety, Childbirth Self-efficacy, and Mode of Delivery in Primiparous Pregnant Women
Acronym: Antenatal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, seyhan Çankaya, Assistant professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201920192019
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Fear of Childbirth; Antenatal Education; Depression, Anxiety; Stress; Childbirth Self Efficacy; Mode of Delivery
Keywords: antenatal education; fear of childbirth; depression; anxiety; stress; childbirth self-efficacy; mode of delivery
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Prior to the study, primiparous pregnant women presented to the outpatient clinic for routine pregnancy control were introduced with free prenatal education classes and they were invited to participate in the study.
  Primiparous women who volunteered to participate in the study and met the inclusion criteria were included in the study and they formed the experimental and control group. Control group did not receive antenatal education and they received prenatal care service routinely provided at the polyclinics of the same hospital.
- Experimental Group (Experimental): Antenatal education group The primiparous pregnant women assigned to the intervention group participated in education classes in groups of 8-10 people. Pregnant women were given structured antenatal education twice a week for two weeks (240 minutes). The total education time was 16 hours. Each session comprised 150 minutes presentation of theoretical knowledge, 45 minutes warm-up and stretching exercises, and 45 minutes relaxation exercises.
  Interventions: Behavioral: Antenat education

INTERVENTIONS:
Behavioral: Antenat education — Antenatal education group The primiparous pregnant women assigned to the intervention group participated in education classes in groups of 8-10 people. Pregnant women were given structured antenatal education twice a week for two weeks (240 minutes). The total education time was 16 hours. Each session comprised 150 minutes presentation of theoretical knowledge, 45 minutes warm-up and stretching exercises, and 45 minutes relaxation exercises.
  Other Names: childbirth preparation training
  Arms: Experimental Group

SUMMARY:
Background: Caesarean delivery rates are quite high, especially in primipara, in Turkey. Fear of birth, low childbirth self-efficacy, and psychological factors may be among the primary causes. Since antenatal educations are not universal and there are differences in educational contents, there is not sufficient evidence on this topic in international studies.

Objective: To investigate the effects of antenatal education on birth fear, depression, anxiety, stress, childbirth self-efficacy, and mode of delivery in primiparous pregnant women.

DETAILED DESCRIPTION:
Background: Caesarean delivery rates are quite high, especially in primipara, in Turkey. Fear of birth, low childbirth self-efficacy, and psychological factors may be among the primary causes. Since antenatal educations are not universal and there are differences in educational contents, there is not sufficient evidence on this topic in international studies.

Objective: To investigate the effects of antenatal education on birth fear, depression, anxiety, stress, childbirth self-efficacy, and mode of delivery in primiparous pregnant women.

Design: A single-blind, prospective, randomized controlled trial. Setting and Participants: The study was conducted in a province in Central Anatolia region in Turkey, and the data were collected between April 2019 and September 2019. Randomized block assignment was used to assign 120 primiparous pregnant women to either the antenatal education group (n = 60) or the control group (n = 60). At the end of the study, 112 women were evaluated.

Measurements: Those in the antenatal education group received two-hour (240 min) educational sessions, twice a week, for 4 weeks. Data were collected by demographic and labor outcomes information form, The Wijma Delivery Expectancy/Experience Questionnaire (Version A and B), Childbirth Self-Efficacy Inventory, and the Depression, Anxiety and Stress Scale.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (between 20 and 32 gestation weeks),
* Healthy,
* Nulliparous with singleton pregnancies,
* Older than 18 years.
* Involved giving birth at full term,
* Having a healthy newborn (born at 38-42 weeks of gestation)

Exclusion Criteria:

* Women taking medication for a diagnosed mental illness (e.g., antidepressants, antianxiety or antipsychotic medication),
* Women with complicated or high- risk pregnancies,
* Anticipating or experiencing a perinatal death (e.g., congenital abnormality incompatible) or stillbirth,
* Having experienced no postnatal complications (hemorrhage, puerperal infection, mastitis, thromboembolic disease or postpartum psychiatric disorder).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ-A) | Change from the Wijma Delivery Expectancy/Experience Questionnaire Version A scores at pre-education and post-education (4 weeks later).
  The W-DEQ Version A was developed by Wijma et al. (1998) in order to measure the fear of childbirth experienced by women during pregnancy. It is a six-point Likert-type scale and consists of 33 items. The responses given to the items on the scale are scored from 0 to 5, where 0 refers to 'extremely' and 5 refers to 'not at all'. The minimum and maximum possible scores to be obtained from the scale are 0 and 165, respectively. As the score increases, so does the fear of childbirth experienced by women (Wijma et al., 1998). Korukcu et al. (2012) examined the validity and reliability of the Turkish version of W-DEQ with women in the last trimester of pregnancy, and found a Cronbach׳s alpha of 0.89 and split-half reliability of 0.91.
Childbirth Self-Efficacy Inventory (CBSEI) | Change from the Childbirth Self-efficacy Inventory scores at pre-education and post-education (4 weeks later).
  The short form of the Childbirth Self-efficacy Inventory has two subscales: outcome expectancy and efficacy expectancy (Ip, et al., 2008). Efficacy expectancy (EE) is a personal conviction about one's ability to successfully perform the required behaviors in a given situation, and outcome expectancy (OE) is the belief that a given behavior will lead to a given outcome. Each subscale consists of 16 items and yields a score between 16 and 160. Higher scores indicate higher levels of efficacy or outcome efficacy for birth. The CBSEI has strong psychometrics, with good internal consistency (α = 0.82) (Ip, et al., 2008). Psychometric properties of the Turkish version of the CBSEI were tested (Ersoy, 2011) and internal consistency was similarly high (α = 0.90).
The depression anxiety and stress scale (DASS-21) | Change from the Depression Anxiety and Stress Scale scores at pre- education, post-education (4 weeks later) and postpartum 6-8 weeks.
  The validity and reliability study of the Depression Anxiety Stress Scale (DASS-21), which was developed by Lovibond and Lovibond (1995), was conducted by Akın and Çetin (2007). The scale consists of 42 items. The scale has a four-point Likert-type rating: (0) Never, (1) Rarely, (2) Frequently, usually, and (4) Always. In the directive of DASS-21, individuals are asked to respond to each item based on how suitable it is for them considering the time period including the previous 30 days. There are 42 items in the DASS-21, 14 of which are related to depression, 14 anxiety, and 14 stress dimensions. The high scores obtained from each of the dimensions of depression, anxiety, and stress indicate that the individual has the relevant problem. The scale has no reverse item and the total score of the scale is expressed between 0 and 42 for each sub-dimension.
The Wijma Delivery Expectancy/Experience Questionnaire B version (W-DEQ-B) | Change from The Wijma Delivery Expectancy/Experience Questionnaire B version (W-DEQ-B) scores at postpartum 6-8 weeks.
  The W-DEQ-B is a 33-item questionnaire with answers based on a 6-point Likert scale. The W-DEQ-B is used to determine fear during childbirth, and feelings and thoughts of postpartum women who had a vaginal childbirth. Total scores can range from 33 to 198, with higher scores indicative of more intense fear of childbirth in the postnatal period. Internal consistency and split-half reliability of the W-DEQ-B are ≥ 0.87 for samples of both nulliparous and multiparous women (Wijma et al., 1998). Reliability and validity studies of the W-DEQ-B were conducted in 2103 in Turkey by Uçar and Beji and the questionnaire's Cronbach's α value was found as 0.88.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Connell MA, Khashan AS, Leahy-Warren P, Stewart F, O'Neill SM. Interventions for fear of childbirth including tocophobia. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013321. doi: 10.1002/14651858.CD013321.pub2. PMID 34231203